CLINICAL TRIAL: NCT04848376
Title: Post-Market Clinical Follow-up Study of A-SPINE's Products
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A-Spine Asia Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: REC108-16
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Degenerative Disc Disease; Kyphosis; Scoliosis; Trauma; Tumor; Stenosis; Pseudoarthrosis of Spine; Deformity
MeSH Terms: conditions — Intervertebral Disc Degeneration; Kyphosis; Scoliosis; Wounds and Injuries; Neoplasms; Constriction, Pathologic; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spine surgery: Use these system:
  (1) SmartLoc (2) SmartLoc Evo(3) Winloc (4) Vigor PEEK Cervical Disc Spacer (5) Combo C (6) Polymer Lumbar Disc Spacer (7) X'Plo (8) Rainboo (9) Combo L
  Interventions: Device: (1) SmartLoc (2) SmartLoc Evo (3) Winloc(4) Vigor PEEK Cervical Disc Spacer (5) Combo C (6) Polymer Lumbar Disc Spacer (7) X'Plo (8) Rainboo (9) Combo L

INTERVENTIONS:
Device: (1) SmartLoc (2) SmartLoc Evo (3) Winloc(4) Vigor PEEK Cervical Disc Spacer (5) Combo C (6) Polymer Lumbar Disc Spacer (7) X'Plo (8) Rainboo (9) Combo L — As long as there are patients using the above device, conduct questionnaire interview.

SUMMARY:
This is a post-market clinical follow-up study that use questionnaires such as Visual Analog Scale (VAS), the Neck Disability Index (NDI), or the Oswestry Disability Index (ODI) to compare the clinical improvement effects before and after surgery.

DETAILED DESCRIPTION:
The purpose of study is to confirm the safety and and performance of the A-SPINE's products for using 2 years. This post-market clinical follow-up study use questionnaires such as Visual Analog Scale (VAS), the Neck Disability Index (NDI), or the Oswestry Disability Index (ODI) to evaluate the clinical improvement effects. Subjects will be evaluated at pre-operation, 6 months, 12 months, and 2 years post treatment. Finally, analyze the clinical outcome, fusion rate, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is above 20 years of age;
* Subject is indicated for A-SPINE Spinal Fixation System;
* Subject is willing and able to provide informed consent to participate in the study;
* Subject is willing and able to understand the purpose of the study, his/her role, and is available to return to the clinic/hospital for all required follow-up visits.

Exclusion Criteria:

* Subjects will be excluded if, in the opinion of the Investigator, the subject does not qualify based on approved labeling requirements or Subject Inclusion Criteria.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients have implanted an A-SPINE device to stabilize the spine and/or restore the height of disc.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-09-08 (Estimated); Study Completion 2022-09-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale- Change from baseline at 2 year | Change from baseline at 2 year
  Visual Analogue Scale is a patient-reported outcome measure. The scale ranges from 0 to 10. A score of 0 represents no pain, while a score of 10 represents extreme pain. Compare baseline and postoperative improvement VAS scores.

SECONDARY OUTCOMES:
Neck Disability Index | Baseline, 6 months, 12 months, 24 months
  The NDI is a questionnaire that is commonly used in clinical trials to measure the self-reported functional status of patients with neck pain.The ten questions are measured on a 6-point scale from 0 (no disability) to 5 (full disability). Compare baseline and postoperative improvement NDI scores.
Oswestry Disability Index | Baseline, 6 months,12 months, 24 months
  The ODI is a questionnaire that is commonly used in clinical trials to measure the self-reported functional status of patients with neck pain.The ten questions are measured on a 6-point scale from 0 (no disability) to 5 (full disability). Compare baseline and postoperative improvement ODI scores.
Number of Device-related Adverse Events | Baseline, 6 months,12 months, 24 months
  Adverse events associated with the device will be assessed at each follow-up visit and the number of cases at the 2-year follow-up will be counted.
Fusion Rate | Baseline, 6 months,12 months, 24 months
  Use X-ray or CT to detect the spine fusion.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Huang, MD, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taichung Tzu Chi Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided